CLINICAL TRIAL: NCT01578785
Title: A Multinational, Multicenter, Randomized, Parallel Group, Double Blind, Placebo Controlled Study Performed in Subjects With Relapsing-Remitting Multiple Sclerosis to Assess the Efficacy, Safety and Tolerability of Glatiramer Acetate 20mg/0.5ml New Formulation Administered Daily by Subcutaneous Injection
Brief Title: An Efficacy, Safety and Tolerability Study of Glatiramer Acetate (GA) 20 mg/0.5 ml New Formulation Administered Daily by Subcutaneous (SC) Injection in Subjects With Relapsing-Remitting Multiple Sclerosis (RRMS)
Acronym: GLOW
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA-MS-302; 2011-005550-57 (EudraCT Number)
Record Dates: First submitted 2012-03-13; First posted 2012-04-17 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-02

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glatiramer Acetate (Experimental): Glatiramer acetate (GA) 20 mg/0.5 ml solution in prefilled syringe for subcutaneous injection once daily.
  Interventions: Drug: Glatiramer Acetate
- Placebo (Placebo Comparator): Placebo solution in prefilled syringe for subcutaneous injection once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glatiramer Acetate — Glatiramer acetate 20mg in 0.5ml for subcutaneous injection in a pre-filled syringe (PFS) is administered daily. Each PFS also contains 20mg mannitol dissolved in water for injection.
  Other Names: Copaxone®
  Arms: Glatiramer Acetate
Drug: Placebo — Matching placebo injection; 20 mg mannitol dissolved in 0.5 mL water for subcutaneous injection in a PFS is administered daily.
  Arms: Placebo

SUMMARY:
This study will investigate the efficacy, safety and tolerability of a new formulation of glatiramer acetate administered at 20 mg/0.5 ml daily versus placebo in patients with Relapsing-Remitting Multiple Sclerosis (RRMS).

DETAILED DESCRIPTION:
Approximately 1400 participants were planned for this study, however only 178 were enrolled prior to early termination.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all inclusion criteria in order to be eligible for the study:

* Subjects must have a confirmed and documented multiple sclerosis (MS) diagnosis as defined by the 2010 Revised McDonald criteria [Ann Neurol 2011: 69:292-302], with a relapsing-remitting disease course.
* Subjects must be ambulatory with a Kurtzke's Expanded Disability Status Scale (EDSS) score of 0-5.5 in both screening and baseline visits.
* Subjects must be in a relapse-free, stable neurological condition and free of corticosteroid treatment [intravenous (IV), intramuscular (IM) and/or by mouth (PO)] or ACTH (adrenocorticotropic hormone) 30 days prior to screening (Month-1) and between screening and baseline (Month 0) visits.
* Subjects must have experienced one of the following:
* At least one documented relapse in the 12 months prior to screening,
* At least two documented relapses in the 24 months prior to screening,
* One documented relapse between 12 and 24 months prior to screening with at least one documented T1-Gd enhancing lesion in a magnetic resonance imaging (MRI) performed within 12 months prior to screening.
* Subjects must be between 18 and 55 years of age, inclusive.
* Women of child-bearing potential must practice an acceptable method of birth control [acceptable methods of birth control in this study include: surgical sterilization, intrauterine devices, oral contraceptive, contraceptive patch, long-acting injectable contraceptive, partner's vasectomy or a double-barrier method (condom or diaphragm with spermicide)].
* Subjects must be able to sign and date a written informed consent prior to entering the study.
* Subjects must be willing and able to comply with the protocol requirements for the duration of the study.

Exclusion Criteria:

Any of the following conditions will exclude the subject from entering the study:

* Subjects with progressive forms of MS.
* Use of experimental or investigational drugs, and/or participation in drug clinical studies within the 6 months prior to screening.
* Use of immunosuppressive agents (including Mitoxantrone and Fingolimod) or cytotoxic agents within 6 months prior to the screening visit.
* Use of natalizumab (Tysabri®) or any other monoclonal antibodies within 2 years prior to screening.
* Use of cladribine within 2 years prior to screening.
* Previous treatment with immunomodulators [including IFNβ 1a and 1b, and IV Immunoglobulin (IVIg)] within 2 months prior to screening.
* Previous use of glatiramer acetate (GA) or any other glatiramoid.
* Chronic (more than 30 consecutive days) systemic (IV, PO or IM) corticosteroid treatment within 6 months prior to screening visit.
* Previous total body irradiation or total lymphoid irradiation.
* Previous stem-cell treatment, autologous bone marrow transplantation or allogenic bone marrow transplantation.
* Pregnancy or breastfeeding.
* Subjects with a clinically significant or unstable medical or surgical condition that would preclude safe and complete study participation, as determined by medical history, physical exams, ECG, abnormal laboratory tests and chest X-ray. Such conditions may include hepatic, renal or metabolic diseases, systemic disease, acute infection, current malignancy or recent history (5 years) of malignancy, major psychiatric disorder, history of drug and/or alcohol abuse and allergies that could be detrimental according to the investigator's judgment.
* A known history of sensitivity to Gadolinium.
* Glomerular filtration rate (GFR) ≤ 60 mL/minute at the screening visit
* Inability to successfully undergo MRI scanning.
* A known drug hypersensitivity to Mannitol.
* Subjects who underwent endovascular treatment for chronic cerebrospinal venous insufficiency (CCSVI).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Boyko, MD, Principal Investigator — Department of Neurology, Russian State Medical University
Locations (169):
- United States (25):
  - Teva Investigational Site 10192, Cullman, Alabama
  - Teva Investigational Site 10204, Fresno, California
  - Teva Investigational Site 10201, La Jolla, California
  - Teva Investigational Site 10196, Centennial, Colorado
  - Teva Investigational Site 10184, Miami, Florida
  - Teva Investigational Site 10180, Sarasota, Florida
  - Teva Investigational Site 10197, Sarasota, Florida
  - Teva Investigational Site 10190, Tampa, Florida
  - Teva Investigational Site 10207, Tampa, Florida
  - Teva Investigational Site 10199, Vero Beach, Florida
  - Teva Investigational Site 10181, Chicago, Illinois
  - Teva Investigational Site 10202, Northbrook, Illinois
  - Teva Investigational Site 10188, Patchogue, New York
  - Teva Investigational Site 10198, Charlotte, North Carolina
  - Teva Investigational Site 10203, Hickory, North Carolina
  - Teva Investigational Site 10209, Hickory, North Carolina
  - Teva Investigational Site 10212, Raleigh, North Carolina
  - Teva Investigational Site 10213, Winston-Salem, North Carolina
  - Teva Investigational Site 10215, Winston-Salem, North Carolina
  - Teva Investigational Site 10194, Akron, Ohio
  - Teva Investigational Site 10191, Dayton, Ohio
  - Teva Investigational Site 10200, Uniontown, Ohio
  - Teva Investigational Site 10206, Cordova, Tennessee
  - Teva Investigational Site 10214, Cordova, Tennessee
  - Teva Investigational Site 10186, Nashville, Tennessee
- Teva Investigational Site 67001, Tirana, Albania
- Belarus (7):
  - Teva Investigational Site 68004, Grodno
  - Teva Investigational Site 68007, Homyel
  - Teva Investigational Site 68003, Minsk
  - Teva Investigational Site 68005, Minsk
  - Teva Investigational Site 68006, Minsk
  - Teva Investigational Site 68001, Vitebsk
  - Teva Investigational Site 68002, Vitebsk
- Bosnia and Herzegovina (4):
  - Teva Investigational Site 69004, Bihać
  - Teva Investigational Site 69002, Mostar
  - Teva Investigational Site 69001, Sarajevo
  - Teva Investigational Site 69003, Tuzla
- Bulgaria (23):
  - Teva Investigational Site 59020, Blagoevgrad
  - Teva Investigational Site 59018, Pleven
  - Teva Investigational Site 59019, Pleven
  - Teva Investigational Site 59025, Pleven
  - Teva Investigational Site 59024, Rousse
  - Teva Investigational Site 59023, Shumen
  - Teva Investigational Site 59006, Sofia
  - Teva Investigational Site 59007, Sofia
  - Teva Investigational Site 59008, Sofia
  - Teva Investigational Site 59009, Sofia
  - Teva Investigational Site 59010, Sofia
  - Teva Investigational Site 59011, Sofia
  - Teva Investigational Site 59012, Sofia
  - Teva Investigational Site 59014, Sofia
  - Teva Investigational Site 59015, Sofia
  - Teva Investigational Site 59016, Sofia
  - Teva Investigational Site 59017, Sofia
  - Teva Investigational Site 59021, Sofia
  - Teva Investigational Site 59026, Sofia
  - Teva Investigational Site 59022, Stara Zagora
  - Teva Investigational Site 59013, Varna
  - Teva Investigational Site 59027, Veliko Tarnovo
  - Teva Investigational Site 59028, Veliko Tarnovo
- Croatia (7):
  - Teva Investigational Site 60003, Osijek
  - Teva Investigational Site 60005, Varaždin
  - Teva Investigational Site 60001, Zagreb
  - Teva Investigational Site 60002, Zagreb
  - Teva Investigational Site 60004, Zagreb
  - Teva Investigational Site 60006, Zagreb
  - Teva Investigational Site 60007, Zagreb
- Estonia (2):
  - Teva Investigational Site 55004, Pärnu
  - Teva Investigational Site 55003, Tallinn
- Georgia (5):
  - Teva Investigational Site 81001, Tbilisi
  - Teva Investigational Site 81002, Tbilisi
  - Teva Investigational Site 81003, Tbilisi
  - Teva Investigational Site 81004, Tbilisi
  - Teva Investigational Site 81005, Tbilisi
- Greece (5):
  - Teva Investigational Site 63017, Athens
  - Teva Investigational Site 63021, Athens
  - Teva Investigational Site 63020, Melíssia
  - Teva Investigational Site 63018, Thessaloniki
  - Teva Investigational Site 63019, Thessaloniki
- Teva Investigational Site 56004, Riga, Latvia
- Mexico (6):
  - Teva Investigational Site 21023, Estado de México
  - Teva Investigational Site 21021, Guadalajara, Jalisco
  - Teva Investigational Site 21022, Mexico City, Distrito Federal
  - Teva Investigational Site 21025, Monterrey
  - Teva Investigational Site 21020, Morelia, Michoacan
  - Teva Investigational Site 21024, San Luís Potosí
- Moldova (4):
  - Teva Investigational Site 70001, Chisinau
  - Teva Investigational Site 70002, Chisinau
  - Teva Investigational Site 70003, Chisinau
  - Teva Investigational Site 70004, Chisinau
- Teva Investigational Site 66001, Podgorica, Montenegro
- North Macedonia (6):
  - Teva Investigational Site 65005, Shtip
  - Teva Investigational Site 65001, Skopje
  - Teva Investigational Site 65002, Skopje
  - Teva Investigational Site 65003, Skopje
  - Teva Investigational Site 65006, Strumica
  - Teva Investigational Site 65004, Tetovo
- Poland (19):
  - Teva Investigational Site 53033, Bialystok
  - Teva Investigational Site 53020, Częstochowa
  - Teva Investigational Site 53023, Gdansk
  - Teva Investigational Site 53024, Gdansk
  - Teva Investigational Site 53031, Grodzisk Mazowiecki
  - Teva Investigational Site 53032, Grodzisk Mazowiecki
  - Teva Investigational Site 53021, Katowice
  - Teva Investigational Site 53019, Kielce
  - Teva Investigational Site 53028, Konstancin-Jeziorna
  - Teva Investigational Site 53037, Kościerzyna
  - Teva Investigational Site 53018, Lodz
  - Teva Investigational Site 53027, Lublin
  - Teva Investigational Site 53036, Olsztyn
  - Teva Investigational Site 53034, Poznan
  - Teva Investigational Site 53030, Poznan / Plewiska
  - Teva Investigational Site 53025, Szczecin
  - Teva Investigational Site 53026, Szczecin
  - Teva Investigational Site 53022, Warsaw
  - Teva Investigational Site 53029, Warsaw
- Romania (12):
  - Teva Investigational Site 52010, Bucharest
  - Teva Investigational Site 52012, Bucharest
  - Teva Investigational Site 52015, Cluj-Napoca
  - Teva Investigational Site 52016, Cluj-Napoca
  - Teva Investigational Site 52017, Constanța
  - Teva Investigational Site 52018, Constanța
  - Teva Investigational Site 52014, Iași
  - Teva Investigational Site 52021, Oradea
  - Teva Investigational Site 52011, Piatra Neamţ
  - Teva Investigational Site 52013, Sibiu
  - Teva Investigational Site 52020, Târgu Mureş
  - Teva Investigational Site 52019, Timișoara
- Russia (23):
  - Teva Investigational Site 50023, Barnaul
  - Teva Investigational Site 50021, Chelyabinsk
  - Teva Investigational Site 50025, Kazan'
  - Teva Investigational Site 50039, Krasnodar
  - Teva Investigational Site 50022, Moscow
  - Teva Investigational Site 50034, Moscow
  - Teva Investigational Site 50035, Moscow
  - Teva Investigational Site 50036, Moscow
  - Teva Investigational Site 50020, Nizhny Novgorod
  - Teva Investigational Site 50024, Nizhny Novgorod
  - Teva Investigational Site 50123, Nizhny Novgorod
  - Teva Investigational Site 50027, Novosibirsk
  - Teva Investigational Site 50019, Perm
  - Teva Investigational Site 50038, Rostov-on-Don
  - Teva Investigational Site 50029, Saint Petersburg
  - Teva Investigational Site 50032, Saint Petersburg
  - Teva Investigational Site 50030, Samara
  - Teva Investigational Site 50037, Saratov
  - Teva Investigational Site 50028, Smolensk
  - Teva Investigational Site 50031, Tyumen
  - Teva Investigational Site 50026, Ufa
  - Teva Investigational Site 50040, Volgograd
  - Teva Investigational Site 50033, Yaroslavl
- Serbia (4):
  - Teva Investigational Site 61002, Belgrade
  - Teva Investigational Site 61005, Belgrade
  - Teva Investigational Site 61001, Kragujevac
  - Teva Investigational Site 61003, Niš
- Ukraine (14):
  - Teva Investigational Site 58022, Chernihiv
  - Teva Investigational Site 58030, Donetsk
  - Teva Investigational Site 58020, Ivano-Frankivsk
  - Teva Investigational Site 58028, Kharkiv
  - Teva Investigational Site 58023, Kyiv
  - Teva Investigational Site 58025, Kyiv
  - Teva Investigational Site 58018, Lviv
  - Teva Investigational Site 58021, Odesa
  - Teva Investigational Site 58029, Poltava
  - Teva Investigational Site 58032, Simferopol, AR Crimea
  - Teva Investigational Site 58031, Uzhhorod
  - Teva Investigational Site 58027, Vinnytsia
  - Teva Investigational Site 58019, Zaporizhzhya
  - Teva Investigational Site 58024, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two hundred seventy-four patients were screened and 178 randomized into the study in a 1:2 treatment arm ratio.
Groups:
- GA 20 MG/0.5 ML: Glatiramer acetate (GA) 20 mg/0.5 ml solution in prefilled syringe for subcutaneous injection once daily.
Period: Overall Study
Arm/Group | Placebo | GA 20 MG/0.5 ML
Started | 59 | 119
Completed | 0 | 0
Not Completed | 59 | 119
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Study terminated by sponsor | 59 | 118

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GA 20 mg/0.5 ml | Total
Number analyzed (Participants) | 59 | 119 | 178
Age, Continuous [Mean (Standard Deviation); unit: years]
  AgeContinuous | 37.7 (9.13) | 38.9 (8.36) | 38.5 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 87 | 132
  Male | 14 | 32 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 59 | 119 | 178
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 58 | 118 | 176
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Bulgaria | 7 | 22 | 29
  Bosnia and Herzegovina | 6 | 11 | 17
  Belarus | 4 | 4 | 8
  Estonia | 0 | 1 | 1
  Georgia | 6 | 8 | 14
  Croatia | 7 | 18 | 25
  Poland | 19 | 35 | 54
  Romania | 9 | 19 | 28
  USA | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Annualized Relapse Rate During the Placebo Controlled Period
Description: The total number of confirmed relapses during the placebo-controlled phase is divided by the sum of the number of days on study in the placebo-controlled phase and then multiplied by the number of days in the year to calculate the annualized relapse rate.
Time Frame: Day 1 up to Month 12
Population: Intent to treat population was planned. However analysis was not performed due to early termination of the study.
Arm/Group | Placebo | GA 20 MG/0.5 ML
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Cumulative Number of New or Enlarging T2 Lesions Measured at Months 6 and 12 (End of Placebo Controlled Period)
Description: Inflammatory disease activity was assessed by magnetic resonance imaging (MRI) measurement of the number of new or newly enlarged T2 lesions.
Time Frame: Day 1 up to Month 12
Population: Intent to treat population was planned. However analysis was not performed due to early termination of the study.
Arm/Group | Placebo | GA 20 MG/0.5 ML
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: The Cumulative Number of Gadolinium-enhancing Lesions on T1-weighted Images Measured at Months 6 and 12 (End of Placebo Controlled Period)
Description: Inflammatory disease activity was assessed by magnetic resonance imaging (MRI) measurement of the number of gadolinium-enhanced T1 lesions.
Time Frame: Day 1 up to Month 12
Population: Intent to treat population was planned. However analysis was not performed due to early termination of the study.
Arm/Group | Placebo | GA 20 MG/0.5 ML
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percent Change From Baseline to Month 12 (End of Placebo Controlled Period) in Brain Volume
Description: Brain atrophy was defined by the percent brain volume change from baseline to Month 12
Time Frame: Day 1 up to Month 12
Population: Intent to treat population was planned. However analysis was not performed due to early termination of the study.
Arm/Group | Placebo | GA 20 MG/0.5 ML
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to day 127
Arm/Group | Placebo | Ga 20 mg/0.5 ml
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/119
Other Adverse Events (participants affected / at risk) | 1/59 | 22/119
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=59) | Ga 20 mg/0.5 ml (N=119)
Injection site erythema (General disorders) | 1 (1) | 13 (13)
Injection site pain (General disorders) | 1 (1) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.